CLINICAL TRIAL: NCT01843569
Title: In Vitro Maturation (IVM) of Human Oocytes
Acronym: IVM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional approval of study has expired.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-364A
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Patients Sensitive to Exogenous Gonadotropins; Ovarian Hyper Stimulation Syndrome (OHSS)
Keywords: In Vitro Maturation; IVM; Natural cycle IVF; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVM (Experimental): All patients registered in this study will undergo natural cycle IVF with In Vitro maturation (IVM) performed on all immature retrieved oocytes.
  Interventions: Biological: In Vitro maturation

INTERVENTIONS:
Biological: In Vitro maturation

SUMMARY:
We hypothesize that the combination of natural cycle IVF or low dose gonadotropin injection combined with In Vitro Maturation (IVM) (Natural IVF/IVM) is a viable option for a selected population of infertility patients who cannot tolerate exogenous gonadotropins or are at risk of ovarian hyperstimulation syndrome.

DETAILED DESCRIPTION:
Natural IVF/IVM may be an attractive treatment alternative to conventional controlled ovarian hyperstimulation (COH)/IVF treatment for infertile women in particular for a select group.

Natural IVF/IVM offers several advantages over conventional COH protocols for IVF including:

1. Elimination of the need for gonadotropin ovarian stimulation
2. Elimination of risk of developing OHSS
3. Simplification of treatment, eliminating the need for frequent blood tests and ultrasound monitoring
4. Reduced cost of treatment
5. Avoiding potential side effects of gonadotropins, including weight gain, bloating, breast tenderness, nausea, mood swings
6. Eliminates concerns about the potential risk of malignancy that may be associated with multiple cycles of ovarian stimulation in a predisposed population.

This pilot study will be conducted to assess the clinical efficacy of natural IVF/IVM

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must be female.
2. Each subject must have an indication for COH and IVF or ICSI.
3. Each subject must be willing and able to provide written informed consent for the trial.
4. Each subject must be ≤42 years of age at the time of signing informed consent.
5. Each subject must have a normal cervical smear result (no atypical or abnormal cells, or in case of atypical squamous or glandular cells, no signs of malignancy; corresponding to Papanicolaou [PAP] I or II) obtained within 12 months prior to signing informed consent must be available.

Exclusion Criteria:

1. Subject with premature ovarian failure.
2. Subject with endocrine abnormalities such as hyperprolactinaemia or thyroid dysfunction.
3. Subject with malformation or absence of uterus.
4. Subject tested positive for Human Immunodeficiency Virus (HIV) or Hepatitis B (by local laboratory; results obtained within 1 year prior to signing ICF are considered valid).
5. Subject with contraindication or allergy/hypersensitivity to hCG, estrogen and progesterone.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 1 month
  Establishment of a successful pregnancy
Implantation | 1 month
  fetal hearts per embryo replaced
live birth rates | 9 months

SECONDARY OUTCOMES:
Multiple pregnancy and miscarriage rates | 9 months
Neonatal outcomes | 9 months
Endocrine parameters (FSH, LH, estradiol [E2], progesterone [P], anti-Mullerian hormone [AMH]) | 2 weeks
Number and size distribution of follicles (≥11 mm, ≥15 mm, and ≥17 mm) as documented by ultrasonography during treatment | 2 weeks
Number and quality of oocytes retrieved | 1 day
Oocyte maturation rate | 1 week
Number of fertilized oocytes | 2 days
Fertilization rate | 1 day
Number and quality of embryos generated | 1 week
Endometrial thickness | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Avner Hershlag, MD, Principal Investigator — NSLIJ
Locations (1):
- The Center for Human Reproduction, Manhasset, New York, United States

REFERENCES:
- [Background] Practice Committee of the American Society for Reproductive Medicine (ASRM). Committee opinion: In Vitro Maturation. Fertil & Steril. Ready for member review 2/21/12. Not yet in print.
- [Background] Le Du A, Kadoch IJ, Bourcigaux N, Doumerc S, Bourrier MC, Chevalier N, Fanchin R, Chian RC, Tachdjian G, Frydman R, Frydman N. In vitro oocyte maturation for the treatment of infertility associated with polycystic ovarian syndrome: the French experience. Hum Reprod. 2005 Feb;20(2):420-4. doi: 10.1093/humrep/deh603. Epub 2004 Nov 4. PMID 15528263
- [Background] Chian RC, Buckett WM, Tan SL. In-vitro maturation of human oocytes. Reprod Biomed Online. 2004 Feb;8(2):148-66. doi: 10.1016/s1472-6483(10)60511-1. PMID 14989791
- [Background] Jurema MW, Nogueira D. In vitro maturation of human oocytes for assisted reproduction. Fertil Steril. 2006 Nov;86(5):1277-91. doi: 10.1016/j.fertnstert.2006.02.126. Epub 2006 Sep 25. PMID 16996508
- [Background] Buckett WM, Chian RC, Holzer H, Dean N, Usher R, Tan SL. Obstetric outcomes and congenital abnormalities after in vitro maturation, in vitro fertilization, and intracytoplasmic sperm injection. Obstet Gynecol. 2007 Oct;110(4):885-91. doi: 10.1097/01.AOG.0000284627.38540.80. PMID 17906024